CLINICAL TRIAL: NCT02853474
Title: Impact of Early Palliative Care on Overall Survival of Patients With Metastatic Upper Gastrointestinal Cancers, Treated With First-line Chemotherapy: a Randomized Phase III Trial
Brief Title: Early Palliative Care in Patients With Metastatic Upper Gastrointestinal Cancers Treated With First-line Chemotherapy
Acronym: EPIC-1511
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Ligue contre le cancer, France (Other); Région Nord-Pas de Calais, France (Other); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EPIC-1511; 2015-A01943-46 (Other: ANSM)
Record Dates: First submitted 2016-07-06; First posted 2016-08-03 (Estimated); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Gastric Cancer; Pancreas Cancer; Bile Duct Cancer; Gastroesophageal Cancer; Esophageal Cancer
MeSH Terms: conditions — Stomach Neoplasms; Pancreatic Neoplasms; Bile Duct Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: Chemotherapy (CT) alone (Sham Comparator): The medical oncologists (or gastro enterologist physician) are in charge of the patient for CT administration, and for the management of symptoms related to the disease and/or the treatment, in accordance with professional practices. If needed (any time), a PC (Palliative consultation) visit could be performed.
  Interventions are :
  * EORTC-QLQ-C30 questionnaire for the assessment of quality of life
  * HADS score for anxiety and depression assessment
  Interventions: Other: EORTC-QLQ-C30 questionnaire; Other: HADS score
- Arm B: CT + Early Palliative care(EPC) (Experimental): Standard oncology care as for arm A plus early PC visits.
  Interventions are :
  * EORTC-QLQ-C30 questionnaire for the assessment of quality of life
  * HADS score for anxiety and depression assessment
  * Early palliative care visits
  Interventions: Behavioral: Early Palliative Care visit; Other: EORTC-QLQ-C30 questionnaire; Other: HADS score

INTERVENTIONS:
Behavioral: Early Palliative Care visit — A PC visit is a visit done by a PC physician. Any kind of visits done by other professionals IS NOT a PC visit.
  Five PC visits are scheduled in this arm.
  Arms: Arm B: CT + Early Palliative care(EPC)
Other: EORTC-QLQ-C30 questionnaire — The Quality of Life is assessed with the QLQ-C30 questionnaire at baseline, 12 and 24 weeks after inclusion, as well as every 8 weeks thereafter.
Other: HADS score — The depression is assessed with the HADS scale (Hospital Anxiety and Depression Scale) at baseline, and then 12 and 24 weeks after inclusion.

SUMMARY:
This prospective, randomized, open-label and multicenter phase III study is aimed to estimate the survival benefit of Early Palliative Care (EPC) combined with standard oncology care including first-line chemotherapy (experimental arm) over standard oncology care only (standard arm), in patients with metastatic upper gastrointestinal cancers (gastric cancer, pancreatic cancer, biliary tract cancers).

DETAILED DESCRIPTION:
Medical oncology is aimed to increase patient's survival, even at metastatic stages, in addition to disease-related and treatment-related symptoms. However, providing palliative care (PC) which includes symptoms management, nutritional support, psychosocial support, as well as assistance on end-of-life preferences, may be as important as survival issues to improve quality of life in such setting. In France, PC has been traditionally offered late, at end-life stage, although the World Health Organization recommends providing PC as earlier as possible in the course of the disease, in order to increase quality of life.

Decades ago, PC services were initiated in France in order to provide a medical alternative to the use of questionable medical practices regarding the end of life period: abandonment, euthanasia, and inappropriate aggressive therapy. According to the French society of palliative care, PC is an approach aimed to provide active care, in a holistic approach, to the person with a serious, progressive or terminal illness. The objective of PC is to relieve pain and other distressing symptoms, but also to take into account the psychological, social and spiritual suffering. PC offers an interdisciplinary support system to help patients and their relatives. As mentioned previously, PC has been in France (but also in the US) usually offered late, at end-life stage. Actually, PC access became a Right guaranteed by the Law, for patients and their families in 1999. This context should explain why even nowadays, PC often means " end of life " not only for the lay-man for the general public but also for caregivers, and some doctors.

The last World Health Organization (WHO) recommendations are far less restrictive than the 1996 French recommendations, as it is stated that PC should be offered as earlier as possible in the course of the disease, in order to increase quality of life, and to positively influence the course of illness. The World Health Organization recommendations add that PC is applicable early in the course of illness, in conjunction with other therapies that are intended to prolong life, such as chemotherapy or radiation therapy, and includes those investigations needed to better understand and manage distressing clinical complications.

In a recent randomized study, 151 patients with newly diagnosed metastatic non-small-cell lung cancer were randomized to receive either early PC (EPC) combined with standard oncologic care or standard oncologic care alone. It was hypothesized that patients, who received EPC, compared with patients who received standard oncologic care only, would have a better quality of life (primary endpoint). The first visit with the PC service set up within the first 12 weeks, and the median number of visits in the EPC group was 4. In this study, the authors referred to the recommendations of the National Consensus Project for Quality Palliative Care. Among patients with metastatic non-small-cell lung cancer, EPC led to significant improvements in quality of life. In addition, EPC led to significant improvements in mood, as well as in overall survival (median survival, 11.6 vs. 8.9 months; HR=0.60, p = 0.02)), despite less aggressive end-of-life care.

Following the publication of this American study, the American Society of Clinical Oncology recommends nowadays that "combined standard oncology care and PC should be considered earlier in the course of the illness for any patient with metastatic cancer….". However, it is clear that a gap exists (not only in France) between this recommendation and the current practice. In addition, there is no consensus on how early PC should be integrated in oncologic services, even though an underpowered small randomized trial reported recently an insignificant better survival favoring early versus delayed (3 months later) initiation of PC.

The results of the study described above, although formally restricted to the field of metastatic non-small-cell lung cancers, have modified the perception of many oncologists about the objectives of PC. However, additional clinical studies should be done before considering EPC as an additional survival input in other advanced malignancies.

The median survival of metastatic upper gastrointestinal (GI) cancers such as pancreatic cancers, gastric cancers, and biliary tract cancers did not exceed 10-11 months, which is as poor as reported with metastatic lung cancers. Standard of care in the metastatic setting in upper GI cancers are described in ad hoc French guidelines, i.e.: "Thésaurus National de Cancérologie Digestive". Briefly, standard of care in metastatic pancreatic cancer in the first-line setting lies on the combination of fluorouracil, irinotecan, and oxaliplatin (FOLFIRINOX regimen) for patients without any cholestasis and in good performance status, and on gemcitabine monotherapy. In metastatic biliary tract cancers, standard of care lies on gemcitabine-based regimen (gemcitabine monotherapy, gemcitabine plus cisplatin, or gemcitabine plus fluorouracil). Besides HER2 positive metastatic gastric/gastrooesophageal patients who present with much better prognosis, and should be treated with trastuzumab-based regimen, most of patients with metastatic gastric/gastrooesophageal HER2 negative patients (IHC + or IHC ++ with negative fish/sish) have poor prognosis, with similar survival rates than patients with other upper GI malignancies. In that setting, several regimens may be offered to patients, such as the following: Folfox, EOX/ECX, Folfiri, LV5FU2-cisplatin, Capecitabine-platinum salt or docetaxel-based regimen ...). Several experimental treatments (antiangiogenics, met inhibitors, modulators of immune check points, etc...) are currently tested in metastatic gastric/gastrooesophageal cancers, but these treatments are restricted to patients in good health condition who accept to participate to clinical trials, and none of these trials have yet produced meaningful survival benefit in the first-line setting.

To summarize, therapeutic advances in the setting of metastatic upper GI cancers are infrequent, and often modest. Providing an extra survival benefit for these patients with EPC, may contribute to deeply modify the practice of care of oncology in France.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an upper gastrointestinal metastatic cancer: pancreatic, biliary tract, esophageal or gastric (including junctional Siewert 2 and 3 cancers) cancers.

NB: gastrooesophageal junctional cancers with dysphagia and/or gastric/gastrooesophageal cancers with unknown or positive HER2 status are not eligible.

* Patients planed to be treated with first-line chemotherapy for metastatic disease.
* Age ≥ 18 years
* Life expectancy ≥ 1 month
* Performance status (OMS) ≤ 2
* Good understanding of French language
* Signed and dated informed consent
* Patients covered by government health insurance

Exclusion Criteria:

* Locally advanced cancer
* Junctional Siewert 1 gastrooesophageal cancer
* Gastric or junctional gastrooesophageal cancer with dysphagia (Atkinson>2)
* Gastric or junctional gastrooesophageal cancer with unknown or positive HER2 status (IHC: +++ or IHC ++ and FISH/SISH +)
* Compression of the biliary tract requiring a bypass

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Overall survival (as intent-to treat analysis) | An average of 1 year
  The overall survival is defined as the time between the date of randomization and the date of death, whatever the cause.

SECONDARY OUTCOMES:
Overall survival (per protocol analysis) | An average of 1 year
  Overall survival curves in per protocol analysis will be given.
One year survival rate (intent-to treat and per protocol analyses) | 1 year
  One year survival rates with their 95% confidence interval in both intent-to-treat and per protocol analyses
Quality of life assessed with the QLQ-C30 | every 8 weeks until the patient withdrawal from the study (during an average of 1 year)
  The Quality of Life is assessed with the QLQ-C30 questionnaire at baseline, and after inclusion, every 8 weeks until patient withdrawal from the study.
Depression assessed with the HADS score | every 8 weeks during 24 weeks
  The depression is assessed with the HADS scale (Hospital Anxiety and Depression Scale) at baseline, and after inclusion, every 8 weeks during 24 weeks.
TUDD (Time Until Definitive Deterioration) | An average of 1 year
  TUDD for Quality of Life scores was defined as the time from randomization to the first observation of a definitive deterioration of QLQ-C30 score or death.
Presence or lack of advanced directives | through study completion, an average of 1 year
  The number of patients whom advanced directives are written in their medical records will be recorded.
Questionnaire "content of PC visits" | during the 6 first months after randomization
  A PC visit is a visit done by a PC physician. Any kind of visits done by other professionals (i.e: dieticians, nurses, social workers, psychologists, pain specialists, etc.) IS NOT a PC visit.
  In Arm B (interventional arm), the content of each PC visit will be described by the PC physician at the end of the visit, by filling a specific check-list built by an ad hoc working-group of PC physicians.
Number of patients treated with chemotherapy | 30 days before death of the patient
  The number of patients treated with chemotherapy in their 30 last days before death will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Arlette Da Silva, MD, Principal Investigator — Centre Oscar Lambret; Antoine Adenis, MD, PhD, Principal Investigator — Centre Oscar Lambret
Locations (20):
- France (20):
  - Institut de cancérologie de l'Ouest-site PAUL, Angers
  - CH de Béthune, Beuvry
  - Centre Hospitalier Boulogne sur Mer, Boulogne-sur-Mer
  - Centre François Baclesse, Caen, Caen
  - Centre Georges Francois Leclerc de DIJON, Dijon
  - Centre Oscar Lambret, Lille
  - Hôpital Saint Vincent de Paul, Lille
  - CHRU, Hôpital Claude HURIEZ, Lille
  - Centre Léon Bérard de LYON, Lyon
  - Institut Paoli-Calmettes de MARSEILLE, Marseille
  - Institut du Cancer de Montpellier, Montpellier
  - Institut de cancérologie de Lorraine, Nancy, Nancy
  - Institut de cancérologie de l'Ouest, Nantes, Nantes
  - Centre Antoine LACASSAGNE DE NICE, Nice
  - Institut Curie, site de Saint Cloud, Hopital, Saint-Cloud
  - CHU de Nantes, CHU - hôpital Nord Laennec,, Saint-Herblain
  - Centre Hospitalier Universitaire de STRASBOURG, Strasbourg
  - Centre Paul Strauss, Strasbourg, Strasbourg
  - Centre Hospitalier de Tourcoing, Tourcoing
  - Centre Hospitalier de Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adenis A, Da Silva A, Ben Abdelghani M, Bourgeois V, Bogart E, Turpin A, Evin A, Proux A, Galais MP, Jaraudias C, Quintin J, Bouquet G, Samalin E, Bremaud N, Javed S, Henry A, Kurtz JE, Cornuault-Foubert D, Vandamme H, Lucchi E, Pannier D, Belletier C, Paul M, Touzet L, Penel N, Chvetzoff G, Le Deley MC. Early palliative care and overall survival in patients with metastatic upper gastrointestinal cancers (EPIC): a multicentre, open-label, randomised controlled phase 3 trial. EClinicalMedicine. 2024 Jun 28;74:102470. doi: 10.1016/j.eclinm.2024.102470. eCollection 2024 Aug. PMID 39526177
- [Derived] Hutt E, Da Silva A, Bogart E, Le Lay-Diomande S, Pannier D, Delaine-Clisant S, Le Deley MC, Adenis A. Impact of early palliative care on overall survival of patients with metastatic upper gastrointestinal cancers treated with first-line chemotherapy: a randomised phase III trial. BMJ Open. 2018 Jan 23;8(1):e015904. doi: 10.1136/bmjopen-2017-015904. PMID 29362244